CLINICAL TRIAL: NCT06064279
Title: Harnessing Allo-immunity to Enhance Immune Checkpoint Inhibitor Responses in Advanced NSCLC
Acronym: HAITEN-ICI
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The funding for this trial was removed.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oncovir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPLP-002-23S; CSR&D (Other Grant/Funding Number: VAMC)
Record Dates: First submitted 2023-09-01; First posted 2023-10-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stage IV NSCLC
Keywords: NSCLC, Immune Checkpoint inhibitor , PDL-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — poly ICLC; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Poly-ICLC + IVIG (Experimental): Patients with stage IV NSCLC will be treated with poly-ICLC + IVIG
  Interventions: Drug: Poly ICLC; Drug: IVIG

INTERVENTIONS:
Drug: Poly ICLC — Tol like receptor 3 agonist
  Other Names: Hiltonol
Drug: IVIG — pooled IVIG

SUMMARY:
Veterans with advanced lung cancer may benefit from recent advances in technologies that is designed to change the activities of their own white blood cells and help kill tumors. However, many cancers can hide from white blood cells making white blood cells less effective in killing tumors. In this study the investigators plan to boost the activity of patients white blood cell by making tumor cells more visible to the white blood cells. This will be done by injecting antibodies and a new drug that together can make white blood cells inside tumors more active. The investigators plan to recruit sixteen people with advanced lung cancer to make sure that this treatment, which has not been done in any humans, is safe and well tolerated.

DETAILED DESCRIPTION:
This is a phase 1b, a first-in-humans, study to examine the safety and feasibility of administration of intratumor (IT) IVIG + poly-ICLC (Hiltonoll®), and intramuscular (IM) poly-ICLC (Hiltonoll®) for the treatment of advanced non-small cell lung cancer (NSCLC) in Veterans without targetable mutations. The investigators will employ the Bayesian optimal interval (BOIN) design 1, with dose escalation, de-escalation endpoints to find the maximum tolerated dose (MTD) in IT injections (IVIG + poly-ICLC) and IM poly-ICLC in 16 subjects while receiving front line Immune Checkpoint inhibitors (ICIs) as the standard of care (SOC). All patients continue to receive ICIs. If safe, a future phase II randomized-controlled study will be designed to determine if treatment with IT injections (IVIG + poly-ICLC) and IM injections (poly-ICLC) results in improved progression free survival.

Primary Objective: To evaluate the safety and determine the MTD as assessed by Common Terminology Criteria for Adverse Events version 6 (CTCAE v. 6) of IT injection of IVIG + poly-ICLC, and IM poly-ICLC given in combination with ICI in Veterans with stage IV NSCLC.

Secondary Objective: To quantitate systemic and tissue-specific immune responses in patients who receive intertumoral IVIG + poly-ICLC, and IM poly-ICLC while receiving ICIs.

Primary Endpoint: Assessment of an MTD dose for IT injection of IVIG + poly-ICLC, and IM injection of poly-ICLC given in combination with ICI in patients with stage IV NSCLC. The primary safety endpoint includes short term and long-term dose limiting toxicity (DLT), and observing less than 25% grade 3 toxicity.

Secondary Endpoints: 1) To assess the correlation of pre-therapy tumor PD-L1 expression with clinical benefit - All tumors will be assessed for PD-L1 expression prior to therapy initiation. 2) To determine the pre-treatment tumor immune infiltrate, and post treatment T cell activation, and correlation with treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with advanced (stage IV) NSCLC
* Eligible to receive ICI/antiPD-1mAb
* No known mutation actionable for first line treatment
* An Eastern Cooperative Oncology Group (ECOG) performance-status (PS) score of 2 or less (ECOG PS is a 5-point scale in which higher scores reflect greater disability)

  * Veterans' responses will be defined as eligible to enroll in HAITEN-ICIs if they meet all criteria
  * To minimize the effects of immunosuppression on the ability to induce antitumor immunity, the investigators will recruit those who have not received systemic cytotoxic chemotherapy (e.g., platinum, taxane, pemetrexed, etc.), do not have major immunosuppression, and are not recipients of organ transplantation
  * Based on our patient population at the MEDVAMC, the investigators estimate that ~30-40% of participants would be receiving systemic chemotherapy and ICIs concurrently, and ~60-70% will be receiving ICI monotherapy
  * Therefore, the investigators anticipate no difficulty in meeting the recruitment goal of 16 persons at our center over two years and ~18 at each of the other sites over the 4-year study period

Exclusion Criteria:

Veterans with

* Concurrent other malignancies, except for localized prostate or localized skin cancer
* Uncontrolled rheumatologic diseases (such as rheumatoid arthritis)
* Current usage of biologics or immunosuppressive therapies
* Status post organ transplant
* An acute respiratory illness (pneumonia, bronchitis, upper respiratory tract infection) in the preceding 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Assessment of an MTD dose for IT injection of IVIG + poly-ICLC, and IM injection of poly-ICLC given in combination with ICI in patients with stage IV NSCLC. The primary safety endpoint includes short term and long-term dose limiting toxicity (DLT), and o | Ten months
  Evaluate the safety as assessed by Common Terminology Criteria for Adverse Events version 6 (CTCAE v. 6) of IT injection of IVIG + poly-ICLC, and IM poly-ICLC given in combination with ICI in Veterans with stage IV NSCLC.

SECONDARY OUTCOMES:
To assess the percent of patients with increase PD-L1 expression and assess clinical outcome after treatment | Ten months
  To quantitate systemic immune responses in patients who receive intratumor IVIG + poly-ICLC, and IM poly-ICLC while receiving ICIs. Pt's adaptive immune cells (T cells) will be examined for the expression of activation markers before and after treatment. The correlation between % changes in immune cell activation and disease progression will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Farrah Kheradmand, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code